CLINICAL TRIAL: NCT03308357
Title: Comparison of the Performance of SB2-Infliximab With Originator Infliximab in the Measure of Serum Concentrations in Serum
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Alfred (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Mark Ward, Dr, The Alfred
Other Study IDs: MSD IIS-57047- GIBSON
Record Dates: First submitted 2017-10-09; First posted 2017-10-12 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Inflammatory Bowel Diseases
Keywords: drug monitoring
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All six subjects: 2 patients with ulcerative colitis; one with active disease and one in remission. 2 patients with Crohn's disease; one with active disease and one in remission. 2 healthly controls. Single blood sample from each participant, serum collected, that serum will be spiked with known concentrations of the originator infliximab and the biosimilar infliximab and then run on a range of assays to measure infliximab drug concentrations
  Interventions: Diagnostic Test: Drug assays to measure infliximab

INTERVENTIONS:
Diagnostic Test: Drug assays to measure infliximab — See protocol

SUMMARY:
The measurement of serum concentrations of infliximab (IFX)has now become a routine part of optimal use of that drug. Trough values are used in two situations: (a) reactively where there is loss of response to infliximab - therapeutic concentrations are indicate likely non-response to the drug, whereas low levels are associated with the chance of regaining response by increasing dosage; or (b) proactively, where dose optimisation in the maintenance phase is performed to ensure ongoing efficacy and/or cost-effective use (where high levels lead to reduction in dosage without loss of efficacy).

With the introduction of biosimilar infliximab into clinical practice, it is important to demonstrate that the biosimilar behaves similarly in the assay used as does originator infliximab to which the assays were developed. While unlikely to be different due to identical protein core, such confirmation is needed before such assays can be used in clinical practice with confidence.

AIMS

1. To compare the concentrations of biosimilar IFX (MSD-IFX) with that of originator IFX (orig-IFX) when added to serum form healthy subjects and those with IBD when measured by commonly-used commercial assays.
2. To compare the effect of freeze-thawing and storage at 4 oC on concentrations of MSD-IFX.

DETAILED DESCRIPTION:
EXPERIMENTAL PLAN Serum This will separated from peripheral blood taken from 2 healthy subjects, 2 patients with ulcerative colitis (one with quiescent and the other with active disease), and 2 patients with Crohn's disease (one with quiescent and the other with active disease). It will be used wither fresh or freshly thawed from serum stored at -20 oC.

Infliximab

Two sources of infliximab will be used:

* Orig-IFX from Janssen
* MSD-IFX from Merck Sharp & Dome.

Preparation of simulated serum samples Fresh or thawed serum will be spiked with IFX to obtained serum at concentrations of 0, 1, 2, 4, 6, 8, 10, 12, 15 and 20 ug/ml. This range covers that seen in routine practice. These preparations will be used fresh or stored in aliquots at 4 oC or -20 oC.

Assays to be evaluated These commercially-available assay kits have been chosen on the basis that they are commonly used. They will all be used according to manufacturer's recommendations.

* SHIKARI Q-INFLIXI from Matriks Biotech;
* LISA TRACKER Premium from Theradiag;
* Promonitor ELISA kit from Grifols;
* Quantum Blue Infliximab trough level rapid test from Buhlmann. Testing protocol The two IFX molecules will be tested on the same plates in duplicate at the concentrations prepared (as above). One assay plate will be sufficient for sera from 2 individuals. One assay only will be performed on any one day.

For the direct comparisons, 3 ELISA assay kits will be required to assess 6 pairs of IFX-spiked sera. The rapid test will be performed in duplicate in a similar way.

In order to assess the effect of storing at -20 oC followed by freeze-thawing, and storage at 4 oC, sera from two subjects will be prepared at one concentration (7 ug/ml), will tested fresh and then again 7 days later after storage at the two temperatures. This will l be performed with one assay kit only (the one performing the best in the comparative studies if differences in kits emerge).

Analysis The result of MSD-IFX will be compared to those of Orig-IFX by plotting the respective curves of concentrations and visually comparing them for each assay. The percent deviation for each concentration will be calculated. The results will also be compared across assays for each IFX source and then the findings compared.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease and ulcerative colitis, deemed to be in remission or with active disease according to validated clinical scoring indices
* healthy controls
* Adult patients able to give informed consent to participate

Exclusion Criteria:

* not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending the inflammatory bowel disease outpatient clinics at Alfred Health. Healthy controls will be doctors attending the clinic
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Drug levels of infliximab originator and biosimilar infliximab | Over the study duration (6 months)
  Infliximab drug levels will be measured on a range of commercially available drug assays

IPD SHARING:
Plan to Share IPD: No